CLINICAL TRIAL: NCT00874926
Title: Efficacy and Safety of Long-term Treatment With KOGENATE Bayer/FS
Brief Title: EFFEKT - Efficacy and Safety of Long-term Treatment With KOGENATE Bayer/FS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 13405; KG0702 (Other: company internal)
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Hemophilia A
Keywords: Octocog alfa; Haemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; F8 protein, human; BAY 14-2222

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Biological: Recombinant Factor VIII (Kogenate FS, BAY14-2222)

INTERVENTIONS:
Biological: Recombinant Factor VIII (Kogenate FS, BAY14-2222) — Haemophilia A patients

SUMMARY:
The aim of this international prospective, non-interventional post-marketing surveillance study is to obtain data on treatment procedures, long-term safety and efficacy and patient acceptance of KOGENATE Bayer in treatment of patients with haemophilia A under daily-life treatment conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of haemophilia A, treated with KOGENATE Bayer/FS as their only source of FVIII, decision taken by the investigator to administer KOGENATE Bayer/FS. For pretreated patients with more than 100 exposure days an inhibitor assessment within three months prior to enrollment should be available; for pretreated patients with less than 100 exposure days an inhibitor assessment at baseline should be available.

Exclusion Criteria:

* Exclusion criteria must be read in conjunction with the local product information.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Haemophilia A patients, no specific study population
Sampling Method: Non-Probability Sample
Enrollment: 405 (Actual)
Dates: Start 2008-06; Primary Completion 2012-11 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Efficacy and Safety of Kogenate Bayer/FS | After 12 months, after 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (17):
- Many Locations, Bahrain
- Many Locations, Bosnia and Herzegovina
- Many Locations, Croatia
- Many Locations, Germany
- Many Locations, Israel
- Many Locations, Kazakhstan
- Many Locations, Kuwait
- Many Locations, Libya
- Many Locations, Morocco
- Many Locations, Oman
- Many Locations, Qatar
- Many Locations, Romania
- Many Locations, Russia
- Many Locations, Saudi Arabia
- Many Locations, Slovenia
- Many Locations, Tunisia
- Many Locations, United Arab Emirates